CLINICAL TRIAL: NCT04932486
Title: Randomised Controlled Trial of Transcutaneous Electrical Stimulation in Obstructive Sleep Apnea
Brief Title: Transcutaneous Electrical Stimulation in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunrise (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7072020000095
Record Dates: First submitted 2021-06-03; First posted 2021-06-21 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous electrical stimulation (Experimental): Participants will be asked to use the stimulator for 6 weeks at home. The study objectives will be evaluated after 6 weeks post-activation of the device.
  Interventions: Device: Transcutaneous electrical stimulation

INTERVENTIONS:
Device: Transcutaneous electrical stimulation — Transcutaneous electrical stimulation of the upper airway muscles

SUMMARY:
The aim of this study is to assess the efficacy of transcutaneous electrical stimulation of the upper airway muscles in patients with obstructive sleep apnea.

ELIGIBILITY:
Inclusion criteria:

* Obstructive apnea-hypopnea index > 15 events/hour
* Patients who do not tolerate or do not accept positive airway pressure therapy

Main exclusion criteria:

* Body mass index < 18.5 or > 32 kg/m2
* Unable or incapable of providing informed written consent
* Unwilling or incapable of returning to all follow-up visits and sleep studies, including evaluation procedures and filling out questionnaires
* Significant co-morbidities making the patient unable or inappropriate to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 6 weeks
  Change from baseline to 6 weeks in the apnea-hypopnea index (AHI)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Benoit Martinot, Principal Investigator — Respisom
Locations (1):
- Respisom, Namur, Belgium